CLINICAL TRIAL: NCT02963051
Title: A Phase Ib Study of Intravenous Copper Loading With Oral Disulfiram in Metastatic, Castration Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopped due to lack of efficacy.
Sponsor: Daniel George, MD (Other)
Collaborators: Give 1 For Dad Campaign (Unknown); The V Foundation for Cancer Research (Other); Peter Michael Foundation (Unknown); Cantex Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Daniel George, MD, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00071007
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Prostate Cancer
Keywords: metastatic castrate-resistant prostate cancer (mCRPC); neuroendocrine prostate cancer (NEPC); adenocarcinoma castrate-resistant prostate cancer (CRPC); Copper; Disulfiram
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Copper; Disulfiram; Gluconates

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Neuroendocrine prostate cancer (NEPC) (Experimental): Subjects with neuroendocrine prostate cancer (NEPC)
  Copper will be administered intravenously at a dose of 1, 3, 5, or 7 mg on cycle 1 days 1, 8, 15. Disulfiram will administered orally at a dose of 80 mg three times a day starting on cycle 1 day 2. Copper gluconate will be administered orally at a dose of 1.5 mg three times a day starting on cycle 1 day 16.
  Interventions: Drug: Copper; Drug: Disulfiram; Drug: Copper gluconate
- Adenocarcinoma CRPC with non-liver/peritoneal metastases (Experimental): Subjects with adenocarcinoma CRPC with non-liver/peritoneal metastases (lymph nodes, bone, or lung)
  Copper will be administered intravenously at a dose of 1, 3, 5, or 7 mg on cycle 1 days 1, 8, 15. Disulfiram will administered orally at a dose of 80 mg three times a day starting on cycle 1 day 2. Copper gluconate will be administered orally at a dose of 1.5 mg three times a day starting on cycle 1 day 16.
  Interventions: Drug: Copper; Drug: Disulfiram; Drug: Copper gluconate
- Adenocarcinoma CRPC with liver and/or peritoneal mets (Experimental): Subjects with adenocarcinoma CRPC with liver and/or peritoneal metastases
  Copper will be administered intravenously at a dose of 1, 3, 5, or 7 mg on cycle 1 days 1, 8, 15. Disulfiram will administered orally at a dose of 80 mg three times a day starting on cycle 1 day 2. Copper gluconate will be administered orally at a dose of 1.5 mg three times a day starting on cycle 1 day 16.
  Interventions: Drug: Copper; Drug: Disulfiram; Drug: Copper gluconate

INTERVENTIONS:
Drug: Copper — 1 mg, 3 mg, 5 mg or 7 mg intravenously on cycle 1 day 1, 8 and 15
  Other Names: Copper chloride
Drug: Disulfiram — 80 mg three times a day
  Source of disulfiram: Cantex Pharmaceuticals
  Other Names: Anatabuse
Drug: Copper gluconate — 1.5 mg three times a day
  Source of copper gluconate: Cantex Pharmaceuticals

SUMMARY:
The purpose of this study is to determine the safety and optimal dosing of intravenous copper chloride and disulfiram in men with metastatic castrate-resistant prostate cancer (CRPC). Eligible men will have neuroendocrine prostate cancer (NEPC), adenocarcinoma CRPC with non-liver/peritoneal metastases (lymph nodes, bone, or lung) or adenocarcinoma CRPC with liver and/or peritoneal metastases. Subjects will receive three doses of intravenous copper chloride and take disulfiram and oral copper gluconate until disease progression (up to two years). Subjects will also undergo a PET scan with radioactive copper 64 to measure the levels of copper in their tumor. The central hypotheses of this project are that (a) copper chloride and disulfiram are safe to give together and that (b) the combination of disulfiram with copper will have efficacy for both mCRPC and NEPC.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Karnofsky performance status ≥ 70
3. Life expectancy of ≥ 12 weeks as determined by treating investigator
4. Adequate laboratory parameters

   * Adequate bone marrow function as shown by: ANC ≥ 1.5 x 109/L, Platelets ≥ 80 x 109/L, Hb>9 g/dL
   * AST/SGOT and ALT/SGPT ≤ 2.5 x Institutional Upper Limit of Normal (ULN)
   * Serum bilirubin ≤ 1.5 x Institutional ULN
   * Serum creatinine ≤ 1.5 x Institutional ULN or 24-hour clearance ≥ 50 mL/min
5. Histologically confirmed diagnosis of prostate cancer. Histologic variants of prostate cancer, including neuroendocrine features and small cell carcinoma of the prostate are included.If neuroendocrine prostate cancer is not biopsy proven, clinical evidence of neuroendocrine prostate cancer is acceptable for stratification into group A.
6. Radiographic evidence of metastatic disease.
7. Ongoing ADT using an LHRH agonist (e.g. leuprolide, goserelin) or antagonist (e.g. degarelix) must continue on therapy unless prior bilateral orchiectomy has been performed. OR Screening serum testosterone must be <50 ng/dl.
8. Evidence of disease progression on ADT as evidenced by one of the following:

   * 2 consecutive PSA levels 50% or greater above the PSA nadir achieved on ADT and separated at least 1 week apart, OR
   * CT or MRI based evidence of disease progression (soft tissue, nodal or visceral disease progression) according to PCWG3 criteria or RECIST 1.1 criteria, or at least 1 new bone scan lesion as compared to the most immediate prior radiologic studies, OR
   * Absolute rise in PSA of 2.0ng/mL or greater, minimum 2 consecutive rising PSA levels with an interval of ≥ 1 week between each PSA level
9. A minimum of 2 weeks elapsed off of antiandrogen therapy prior to registration (i.e. flutamide, nilutamide, and bicalutamide) without evidence of an anti-androgen withdrawal response. An anti-androgen withdrawal response is a PSA level at 2 weeks (or more) off of anti-androgen equal or higher than PSA level when anti-androgen therapy stopped.
10. For subjects in Groups B or C, previous use of at least one androgen pathway inhibitor (either abiraterone acetate or enzalutamide) for metastatic CRPC
11. For subjects in Group A with NEPC, previous use of at least one platinum-containing chemotherapy regimen.
12. A minimum of 2 weeks off of enzalutamide or abiraterone if applicable, prior to registration.
13. A minimum of 4 weeks from prior chemotherapy, including but not limited to, docetaxel, cabazitaxel, mitoxantrone, carboplatinum, cisplatin, or estramustine; if applicable, prior to registration.
14. A minimum of 4 weeks from any major surgery prior to registration.
15. Ability to swallow, retain, and absorb oral medication.
16. Ability to understand and the willingness to sign a written informed consent document.
17. Willingness to abstain from alcohol or any alcohol-containing fluids for the duration of the study.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Symptomatic subjects who accept treatment with approved palliative or life-prolonging systemic therapies, including docetaxel and cabazitaxel chemotherapy. (Note: subjects who refuse chemotherapy or are not symptomatic or in immediate need for standard systemic therapies may be included.)
2. Known history of Wilson's disease or a copper deficiency.
3. Uncontrolled hypertension (systolic BP >160 mmHg or diastolic BP > 95 mmHg) or other medical condition that could jeopardize the assessment of toxicity on study.
4. Active or symptomatic viral hepatitis or chronic liver disease.
5. Known history of Hepatitis B Virus (HBV) or Hepatitis C (HCV) infection.
6. Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class II-IV heart disease or cardiac ejection fraction measurement of < 50% at baseline.
7. Symptomatic atrial fibrillation or other cardiac arrhythmia for which the therapy is not stable or requiring changes in therapy within 1 month of treatment initiation. Atrial fibrillation or other cardiac arrhythmia which is clinically stable on stable therapy is allowed.
8. Corrected QT interval calculated by the Bazett formula (QTcB) >480 msec.
9. Other malignancy, except non-melanoma skin cancer, with a ≥ 30% probability of death within 24 months.
10. Administration of an investigational therapeutic within 30 days of Cycle 1, Day 1.
11. Any condition which, in the opinion of the investigator, would preclude participation in this trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Up to 2 years
  Safety (NCI CTC v4.0) and tolerability of IV CuCl2 and DSF in men with mCRPC

SECONDARY OUTCOMES:
Median radiographic progression free survival (PFS) | Every 12 weeks, up to 2 years
  Radiographic PFS based on PCWG3 criteria or based on the onset of a skeletal related event. Imaging obtained every 12 weeks.
Amount of 64-Copper uptake by the tumor | Baseline
  64-Copper PET imaging
Change in PSA | Every 4 weeks, up to 2 years
  PSA response
Time to PSA nadir | Every 4 weeks, up to 2 years
  Time to PSA nadir
Time to PSA progression | Every 4 weeks, up to 2 years
  Time to PSA progression

CONTACTS AND LOCATIONS:
Overall Officials: Daniel George, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States